CLINICAL TRIAL: NCT06003049
Title: An Investigator-Initiated, Single Center, Prospective, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate Safety and Efficacy of OnabotulinumtoxinA (BOTOX®) in Adults With Moderate Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study to Evaluate Safety and Efficacy of BOTOX in Adults With Moderate COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RMW Testing (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COPD 101
Record Dates: First submitted 2023-08-04; First posted 2023-08-21 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: This is an Investigator-initiated a clinical trial to determine the safety and preliminary efficacy of subcutaneous injections of BOTOX in participants with moderate COPD.
  Participants will be treated with either one series of subcutaneous injections of BOTOX or of normal saline solution in the back in the T-1 to T-5 dermatome regions as indicated in Appendix A.
  Participants' COPD status will be measured using the COPD Assessment Test (CAT), Pulmonary Function Test (Spirometry), and 6 Minute Walk Test (6MWT).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Active Comparator): OnabotulinumtoxinA
  Interventions: Drug: OnabotulinumtoxinA
- Placebo Arm (Placebo Comparator): Normal saline
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: OnabotulinumtoxinA — BOTOX injection series
  Other Names: BOTOX
  Arms: Treatment Arm
Other: Placebo — Placebo injection series
  Arms: Placebo Arm

SUMMARY:
The aim of this clinical trial to determine the safety and effectiveness of treating the COPD symptoms with subcutaneous BOTOX injections in participants with moderate COPD.

DETAILED DESCRIPTION:
This is a prospective, double-blind, randomized, placebo-controlled, investigator-initiated clinical trial to assess the safety, tolerability, and efficacy using an approved drug, BOTOX, in moderate COPD participants.

Forty participants with moderate COPD, defined as mMRC Dyspnea Scale scores of grades 2 or 3 and CAT scores of 12 to 20, will be included. If eligibility criteria are met, subjects will be randomized to either the treatment arm (BOTOX) or placebo, treated on day one and observed for 90 days for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. History of moderate COPD as diagnosed by a physician
3. FEV1 /FVC Ratio < 0.7 with Post-Bronchodilator FEV1 ≥50% of predicted value at Screening
4. Modified Medical Research Council (mMRC) Dyspnea Scale score of Grade 2 or 3 (Appendix B) at Screening
5. CAT score of 12-20 (Appendix C) measured at Screening and confirmed at Baseline
6. Ability to consent
7. Ability to receive subcutaneous injections along the spine/back in the T-1 > T-5 region
8. Females of reproductive potential must have a negative pregnancy test at screening and use of highly effective contraception method (refer to section 12.3.9) for 4 weeks after study drug administration. Women are generally considered to be of reproductive potential if a non-menopausal female has not had a hysterectomy, bilateral oophorectomy, or medically documented ovarian failure.
9. Males of reproductive potential must use condoms with spermicide or other methods to ensure effective contraception with partner for 4 weeks after study drug administration. Men are generally considered to be of reproductive potential if they can produce sperm.

Exclusion Criteria:

1. Any medical condition that may put the participant at increased risk with exposure to botulinum toxin type A (BTX-A), including, but not limited to diagnoses of myasthenia gravis (MG), Eaton-Lambert syndrome, amyotrophic lateral sclerosis, multiple sclerosis, or any other significant disease that might interfere with neuromuscular function
2. Treatment of study target treatment area using acupuncture, transcutaneous electrical stimulation (TENS), cranial traction or injection of anesthetics/steroids within 4 weeks prior to the screening visit (oral or inhaled steroids are allowed)
3. Known allergy to BTX-A
4. Known history of pulmonary hypertension
5. Documented COPD exacerbation within 4 weeks of Baseline (Day 1)
6. Post-bronchodilator FEV1 value ≤30% of the predicted value at screening
7. Current smoker (e-cigarettes or cigarettes, cigars, pipe tobacco, vape)
8. Prior or current lung cancer
9. Post COVID symptoms resulting in breathing difficulties beyond pre-COVID COPD symptoms
10. Allergy to local anesthetics
11. History of botulism
12. Has an active pulmonary infection requiring systemic therapy within 14 days prior to the baseline visit
13. Known/documented medical history of clotting disorders
14. Pregnant or breastfeeding
15. Requires immediate admission to the hospital during screening that would render the participant unable to comply with the protocol
16. Any serious medical condition, such as kidney, liver, or cardiac disease, asthma, angioedema, bleeding disorder, malignancy, seizure, neutropenia, AIDS, that in the judgement of the Investigator could confound study assessments
17. Any condition (physical, mental, or social), occupational reason or other responsibility that, in the judgment of the Investigator, would jeopardize the safety or rights of the study participant, or render the participant unable to comply with the protocol, including participant's return for follow-up visits on schedule
18. Any chronic conditions which may cause diffusion of excess of Substance P in the cerebrospinal fluid (CSF), including but not limited to diabetes, chronic kidney failure, cirrhosis, pancreatitis, osteoporosis, ongoing clinical depression, migraines and fibromyalgia, that would compromise the participant's safety as determined by the Investigator.
19. History of keloid formation after injury.
20. Treatment with another investigational drug or other investigational intervention within 2 weeks of study start and throughout study duration
21. Treatment with any botulinum toxin (BoNT) products within 6 months of the baseline visit.
22. Any abnormal laboratory value greater than 3 times upper limit of normal (ULN) for albumin, total protein, alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase (ALP), and bilirubin), and 5 times the upper limit of normal (ULN) for all other lab values.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
CAT (Average) | 28 days
  The COPD Assessment Test (CAT) is assessed to capture the health status. The total score ranges from 0 to 40 points. Average change in CAT score over 28 days between treatment arms with a higher scores indicating a more significant change in health status.

SECONDARY OUTCOMES:
CAT (Change in Units) | 28 days
  The COPD Assessment Test (CAT) is assessed to capture the health status. The total score ranges from 0 to 40 points. Portion of participants with a change in score of 2 or greater are indicating a change health status between baseline and day 28 follow-up assessment.
FEV1 | 28 days
  Percentage of predicted (% pred) of the forced expiratory volume in 1 second (FEV1). FEV1 values that are ratios that are higher than at baseline suggest an improving health status. Assessment at Baseline and day 28 follow-up assessment
FEV1/FVC | 28 days
  Ratio of percentage of predicted (% pred) of the forced expiratory volume in 1 second to (FEV1ercentage of predicted (% pred) of the forced vital capacity (FVC). FEV1/FVC ratios that are higher than at baseline suggest an improving health status. Assessment at baseline and day 28 follow-up assessment.
6MWT | 28 days
  The six-minute walk test (6MWT) is performed to capture the longest 6MWT for further analyses. The longer distance covered indicates an improving health status. Assessment at baseline and day 28 follow-up assessment.
COPD Exacerbations | 90 days
  Exacerbations of chronic obstructive pulmonary disease (COPD) are episodes of worsening of symptoms, leading to substantial morbidity and mortality. Total number of exacerbations will be analyzed and measured at baseline, all follow-up and end of trial assessments. More exacerbations experienced over time indicate a worse health status.
Adverse Reactions | 90 days
  The number of reported adverse reactions and serious adverse events per participant. The more adverse reactions, the worse the health status of the participant measured at baseline, all follow-up and end of trial assessments.

OTHER OUTCOMES:
CAT Score | 90 days
  The COPD Assessment Test (CAT) is assessed to capture the health status. The total score ranges from 0 to 40 points. Change in CAT score measured at baseline, all follow-up and end of trial assessments between treatment and placebo arms with a higher scores indicating a more significant change in health status.
FEV1 | 90 days
  Percentage of predicted (% pred) of the forced expiratory volume in 1 second (FEV1). Change in FEV1 measured at baseline, all follow-up and end of trial assessments between treatment and placebo arms with a higher scores indicating a more significant change in health status.
FEV1/FVC | 90 days
  Ratio of percentage of predicted (% pred) of the forced expiratory volume in 1 second to (FEV1ercentage of predicted (% pred) of the forced vital capacity (FVC). FEV1/FVC measured at baseline, all follow-up and end of trial assessments between treatment and placebo arms with a higher scores indicating a more significant change in health status.
Vital Signs: Oxygen saturation | 90 days
  Oxygen saturation (SpO2) measured at baseline, all follow-up and end of trial assessments between treatment and placebo arms with a higher scores indicating a more significant change in health status.
6MWT | 90 days
  The six-minute walk test (6MWT) is performed to capture the longest 6MWD for further analyses. 6MWT measured at baseline, all follow-up and end of trial assessments between treatment and placebo arms with a higher scores indicating a more significant change in health status.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Do, Principal Investigator — Investigator
Locations (1):
- Tranquil Clinical Research, Webster, Texas, United States

IPD SHARING:
Plan to Share IPD: No